CLINICAL TRIAL: NCT04301687
Title: The Analgesic Efficacy of the Ultrasound-Guided Femoral Articular Branch Block for Ambulatory Hip Arthroplasty: A Randomized-Controlled Trial Secondary IDs:
Brief Title: FAB Block vs. Placebo for Hip Arthroplasty Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAB for Hip Arthroplasty
Record Dates: First submitted 2020-01-22; First posted 2020-03-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthroplasty; Anesthesia, Regional; Femoral Articular Branch Block

STUDY DESIGN:
Intervention Model Description: Patients will be randomized between one of two treatment groups. The intervention of femoral articular branch block or the control group (non-invasive placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist performing the nerve block will be aware of group allocation; but a separate anesthesiologist providing intra-operative care will remain blinded. The patient and the research staff collecting outcome data will remain blinded until all data are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Articular Branch Block (Experimental): Patients will receive an ultrasound-guided femoral articular branch block with an injection of 20ml of ropivicaine 0.5%
  Interventions: Procedure: Femoral Articular Branch Block
- Placebo Block (Placebo Comparator): Patients will receive an ultrasound simulation of the location of a femoral articular branch block , this is to maintain blinding. A subcutaneous injection of 1ml of normal sterile saline will be administered
  Interventions: Procedure: Placebo Block

INTERVENTIONS:
Procedure: Femoral Articular Branch Block — Slow injection (3mL aliquots) of local anesthetic solution (20ml of Ropivacaine 0.5%) into the fascia above the iliopsoas muscle (located in the groove between the two bony landmarks - (1)anterior inferior iliac crest and (2)iliopubic eminence).This is done by ultrasound guidance.
  Arms: Femoral Articular Branch Block
Procedure: Placebo Block — Subcutaneous injection of 1ml normal sterile saline
  Arms: Placebo Block

SUMMARY:
Hip arthroplasty surgery can be associated with significant pain. A regional anesthesia technique, the femoral articular branch block (FAB), has recently been proposed to collectively block terminal femoral and accessory obturator nerve branches to the hip joint with a single injection, theoretically blocking most of the innervation relevant to hip arthroscopy while sparing the main femoral nerve branches to the quadriceps muscles. The investigators aim to demonstrate the analgesic benefits of FAB. The investigators hypothesize that FAB will reduce opioid consumption and improve postoperative quality of recovery in patients having hip arthroplasty. This is a randomized, controlled, double-blind study and half the patients will be randomized to receive the femoral articular branch block and the other half of patients will be randomized to receive a placebo block. A comparison of pain will be made between both groups.

DETAILED DESCRIPTION:
Hip arthroplasty procedure is frequently associated with severe post-operative pain despite the practice of injecting the hip joint with local anesthetics at the end of the procedure and the use of intraoperative opioids. These patients usually receive a spinal anesthetic as well. The ideal analgesic technique that provides adequate pain relief following this procedure has not been established yet.

The femoral articular branch block (FAB) has recently been proposed to collectively block the terminal femoral and accessory obturator nerve branches to the hip joint with a single injection, theoretically blocking most of the innervation relevant to hip arthroscopy while sparing the main femoral nerve branches to the quadriceps muscle. The investigators aim to demonstrate the analgesic benefits of FAB.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Ages 18-60yrs
* BMI ≤ 35 kg/m2

Exclusion Criteria:

* Preexisting neurological deficits or peripheral neuropathy in the distribution of femoral, obturator, or lateral cutaneous nerves
* Local infection
* Contra-indication to regional anesthesia e.g. bleeding diathesis, coagulopathy
* Chronic pain disorders
* History of use of over 30mg oxycodone or equivalent per day
* Contraindication to a component of multi-modal analgesia
* Allergy to local anesthetics
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy
* Inability to provide informed consent
* Patient refusal of FAB
* Revision arthroscopy surgeries

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Analgesic Consumption | 24 hours postoperatively
  Postoperative cumulative oral morphine equivalent consumption during the first 24 hours will be the first primary outcome
Quality of Life scores | 24 hours postoperatively
  Quality of Recovery (QR15) scores at 24 hours will be the second primary outcome.

SECONDARY OUTCOMES:
Pain Assessment (VAS) | Up to 48 hours post-operatively
  Visual Analogue Scale(VAS) - Pain:Overall pain assessed at rest and on movement A continuous scale comprised of a 100mm (10cm) horizontal line, anchored by 2 verbal descriptions No Pain to Worst Pain
Analgesic Consumption | Up to 48 hours following surgery
  Consumption intra-operatively, total in-hospital postoperative consumption, and time to first analgesic request in the first 24 hours, cumulative oral morphine equivalent
Incidence of block-related complications | Up until one month following nerve block
  vascular puncture, hematoma formation, intravascular injection, epidural anesthesia-bilateral sensory block
Block Success | 4 hours after nerve block has been administered
  Sensory and motor block onset assessment in the 3 nerves involved will be performed every 5 minutes post block procedure up until 30 minutes and then one, two, and four hours postoperatively.
Patient Satisfaction with Analgesic Technique | One month after surgery
  A Patient Diary will be completed to assess overall satisfaction with analgesic technique
Demographic Data | Day 1 - first 24 hours
  Patient demographics - There is no scale, just questions asked of the participant.
Incidence of opioid-related side effects | Up until one month following nerve block
  nausea, vomiting, pruritus, sedation

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — Women's College Hospital

IPD SHARING:
Plan to Share IPD: No